CLINICAL TRIAL: NCT00842452
Title: A Phase I Study of Weekly Oral Topotecan in Gynecologic Malignancies
Brief Title: Topotecan in Treating Patients With Gynecologic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Steven Waggoner, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Steven Waggoner, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Y08; P30CA043703 (NIH); CASE2Y08 (Other: Case Comprehensive Cancer Center); CASE 2Y08-CC630 (Other: Cancer Center IRB); NCI-2009-01290 (Registry Identifier: NCI)
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Sarcoma; Vaginal Cancer; Vulvar Cancer
Keywords: recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent vaginal cancer; stage III vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent vulvar cancer; stage III vulvar cancer; stage IV vulvar cancer; recurrent cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; fallopian tube cancer; ovarian sarcoma; ovarian stromal cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Sarcoma; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Topotecan (Experimental)
  Interventions: Drug: topotecan hydrochloride; Other: pharmacological study

INTERVENTIONS:
Drug: topotecan hydrochloride — Patients receive oral topotecan hydrochloride on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Other: pharmacological study — Patients treated at the maximum tolerated dose undergo blood sample collection periodically on day 1 of course 1 for pharmacokinetic studies.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of topotecan in treating patients with gynecologic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum tolerated dose (MTD) of oral topotecan hydrochloride in patients with unresectable gynecologic malignancies.
* To determine the safety and tolerability of this drug in these patients.
* To obtain pharmacokinetic data to assess plasma concentrations of this drug when administered at the MTD.

Secondary

* To explore the response in patients treated with this drug.

OUTLINE: Patients receive oral topotecan hydrochloride on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients treated at the maximum tolerated dose undergo blood sample collection periodically on day 1 of course 1 for pharmacokinetic studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or cytologically confirmed unresectable gynecologic malignancy for which standard curative or palliative care is not available

  * All tumor types allowed NOTE: *Histologic confirmation of recurrence is not required
* Measurable or nonmeasurable disease

  * If CT scan was used to evaluate measurable disease, lesions must be clearly defined and be ≥ 10 mm on spiral CT scan
* No "borderline tumors" or tumors with low malignant potential

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 60 mL/min
* AST/ALT ≤ 2.5 times ULN (< 5 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 2.5 times ULN (< 5 times ULN if liver metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate intestinal function (i.e., no gastrostomy tube or requirement for IV hydration or nutritional support)
* No severe gastrointestinal bleeding or intestinal obstruction
* No other condition that would affect gastrointestinal absorption and motility
* No septicemia, severe infection, or acute hepatitis
* No other malignancies requiring chemotherapy or radiotherapy within the past 5 years, except skin cancer
* No concurrent severe medical problem unrelated to the malignancy that would significantly limit full compliance with the study, expose the patient to extreme risk, or decrease life expectancy

PRIOR CONCURRENT THERAPY:

* At least 28 days since prior investigational drugs (including cytotoxic drugs)
* At least 4 weeks since prior chemotherapy, radiotherapy, biologic therapy, or surgery and recovered
* No more than 3 prior chemotherapy regimens
* No prior topotecan hydrochloride or other camptothecin analogs
* No prior radiotherapy to > 25% of the bone marrow
* No other concurrent chemotherapy, radiotherapy, biologic therapy, immunotherapy, or hormonal therapy for cancer
* No concurrent administration of any of the following:

  * P-glycoprotein (ABCB1, Pgp, MDR1) inhibitors or inducers
  * Breast cancer-resistant protein (ABCG2, BCRP, MXR) inhibitors or inducers
* No concurrent chronic H2 antagonists, proton pump inhibitors, or antacids for gastritis, gastroesophageal reflux disease, or gastric or duodenal ulcers

  * Intermittent antacid therapy is allowed provided it is given ≥ 6 hours prior to and ≥ 90 minutes after study drug administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Treatment repeats every 28 days for up to 6 courses in the absence of unacceptable toxicity.
Safety and tolerability | Treatment repeats every 28 days for up to 6 courses in the absence of unacceptable toxicity.
Plasma concentration of topotecan hydrochloride when administered at the MTD | blood sample collection periodically on day 1 of course 1 for pharmacokinetic studies

SECONDARY OUTCOMES:
Response | Treatment repeats every 28 days for up to 6 courses in the absence of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Waggoner, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States